CLINICAL TRIAL: NCT00552526
Title: Comparing Ketogenic Diet With the Most Appropriate Antiepileptic Drug- a Randomized Study of Children With Mental Retardation and Drug Resistant Epilepsy
Brief Title: Ketogenic Diet vs.Antiepileptic Drug Treatment in Drug Resistant Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Rikshospitalet-Radiumhospitalet HF (Bjorn Bjurulf), Rikshospitalet-Radiumhospitalet HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ketogenic diet; EudraCT:2006-001776-20
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Epilepsy; Mental Retardation
Keywords: Epilepsy; Children; Mental retardation; Ketogenic diet; Diet
MeSH Terms: conditions — Epilepsy; Intellectual Disability | interventions — Diet, Ketogenic; Anticonvulsants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketogenic diet (Active Comparator)
  Interventions: Dietary Supplement: Ketogenic diet
- AED (Active Comparator): Most appropriate antiepileptic drug
  Interventions: Drug: Antiepileptic drug (AED)

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic diet is a very strict high fat diet
  Arms: Ketogenic diet
Drug: Antiepileptic drug (AED) — An AED,not used by the patient before, which we consider to be the most appropriate will be given orally or by gastrostomy. Serum concentration, the body weight, side effects and effects on the epilepsy will be considered when deciding the dose of the AED. Traditions for amount of medicine/kg body weight or optimal serum concentration at our center will be followed. This tradition will be the same as in other major European epilepsy centers but might propose lower, but not higher amounts than recommended by the drug company. Drugs from ACT groups N03A, N05BA, N05CD, H02A or S01EC will be used including prednisolon,levetiracetam, valproate, carbamazepine, oxcarbazepine, topiramate, felbamate, zonisamide, vigabatrin, tiagabil, lamotrigine, pregabalin, rufinamide, clobazam, clonazepam, tiagabine, gabapentin, phenytoin, phenobarbital, ethosuximide, acetazolamide, nitrazepam and other new antiepileptic drugs that might be released during the study period.
  Arms: AED

SUMMARY:
This is an open randomized controlled study in children with mental retardation and refractory epilepsy in which treatment with ketogenic diet (KD) is compared with treatment with the antiepileptic drug (AED), not tried by the patient before, which we consider to be the most appropriate AED for the patient.

DETAILED DESCRIPTION:
There are two trials in the study:

* To compare the effect of the ketogenic diet with the effect of the most appropriate AED after 4 months
* To evaluate the effect of the ketogenic diet after 4 and 13 months on the children who have been randomized to this treatment, the seizure frequency is compared with the frequency before start of treatment

ELIGIBILITY:
Inclusion Criteria:

* The patient is mentally retarded
* The patient has tried at least 3 different AED:s including one combination with two or more different AED:s.
* The parents are willing to include their child in the study after written and verbal information.
* Patients with all types of epilepsy can be included.
* The patient has at least 6 seizures/month.
* The patient is submitted to our epilepsy center.
* The seizures are possible to count
* The patient has either generalized epilepsy, multifocal epilepsy or an epilepsy where it is undetermined whether it is localized or generalized such as Dravet syndrome classified as G40.3-G40.9 in ICD X.

Exclusion Criteria:

* The family is expected to have compliance problems with treatment and/or seizure registration.
* The hospital which have submitted the patient is not willing to accept the inpatient stays and the procedures that are necessary for the project.
* The patient's seizures are under acceptable control.
* The patient has got a vagus nerve stimulator implanted within the last 18 months, has started a new antiepileptic drug within the last 2 months or has changed his antiepileptic drugs the last month.
* The patient has a medical condition, for example a metabolic disease, where ketogenic diet is contraindicated.
* The patient has a localized epilepsy classified as G40.0-G40.2 in ICD X.
* The patient's nutritional status is not good enough or intake of fluid is to small to permit treatment with ketogenic diet.
* The patient has within the last 2 months been using medications or herbal medications that has a considerable effect on glucose metabolism, such as oral glucocorticoids.
* The patient has within the last 2 months been using medications or herbal medications that has a considerable effect on metabolism of AED:s.
* The patient uses herbal medicine which can interact with AED or Ketogenic diet.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-01 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Comparing amount of patients with 100%, >90% and >50% reduction in number of seizures between the two groups of seizures | 4 months

SECONDARY OUTCOMES:
Comparing the parents´evaluation of change in quality of life and cognitive function between the two groups. The parents will answer a questionary. | Four months
Comparing side effects between the two groups | Four months
Comparing change in slow activity and epileptic activity by template matching on 24 hour EEG | Four months
Investigating side effects and change in number of seizures, change in EEG, quality of life and cognitive function after 13 months of treatment with the ketogenic diet | 13 months
Is the effect of the ketogenic diet as good in children with severe mental retardation as in children with less severe learning disabilities? | 4 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Bjurulf, MD, Principal Investigator — SSE, Nevrological dep., Rikshospitalet University Hospital
Locations (1):
- SSE, Nevrological dep. , Rikshospitalet University hospital, Oslo, Norway

REFERENCES:
- [Background] Pulsifer MB, Gordon JM, Brandt J, Vining EP, Freeman JM. Effects of ketogenic diet on development and behavior: preliminary report of a prospective study. Dev Med Child Neurol. 2001 May;43(5):301-6. doi: 10.1017/s0012162201000573. PMID 11368482
- [Background] Hallböök T Effects of vagus nerve stimulation and ketogenic diet on quality of life and changes in EEG and sleep Lund University 2006
- [Background] Kossoff EH, McGrogan JR. Worldwide use of the ketogenic diet. Epilepsia. 2005 Feb;46(2):280-9. doi: 10.1111/j.0013-9580.2005.42704.x. PMID 15679509
- [Background] Levy R, Cooper P. Ketogenic diet for epilepsy. Cochrane Database Syst Rev. 2003;(3):CD001903. doi: 10.1002/14651858.CD001903. PMID 12917915
- [Background] Kang HC, Kim YJ, Kim DW, Kim HD. Efficacy and safety of the ketogenic diet for intractable childhood epilepsy: Korean multicentric experience. Epilepsia. 2005 Feb;46(2):272-9. doi: 10.1111/j.0013-9580.2005.48504.x. PMID 15679508
- [Background] Kossoff EH, Pyzik PL, McGrogan JR, Vining EP, Freeman JM. Efficacy of the ketogenic diet for infantile spasms. Pediatrics. 2002 May;109(5):780-3. doi: 10.1542/peds.109.5.780. PMID 11986436
- [Background] Lefevre F, Aronson N. Ketogenic diet for the treatment of refractory epilepsy in children: A systematic review of efficacy. Pediatrics. 2000 Apr;105(4):E46. doi: 10.1542/peds.105.4.e46. PMID 10742367